CLINICAL TRIAL: NCT01869517
Title: Myoring Versus Keraring Implantation for Keratoconus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, clinical professor ,ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 91138
Record Dates: First submitted 2013-05-22; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrastromal corneal continuous ring (Myoring) (Active Comparator)
  Interventions: Other: Intrastromal corneal continuous ring (Myoring) implantation
- Intrastromal corneal ring segments (Keraring) (Active Comparator)
  Interventions: Other: intrastromal corneal ring segments (Keraring) implantation

INTERVENTIONS:
Other: intrastromal corneal ring segments (Keraring) implantation
  Arms: Intrastromal corneal ring segments (Keraring)
Other: Intrastromal corneal continuous ring (Myoring) implantation
  Arms: Intrastromal corneal continuous ring (Myoring)

SUMMARY:
Various approaches, including surgical and non-surgical management have been proposed for keratoconus. One of the surgical procedures is Intrastromal Corneal Ring implantations that have been designed to achieve refractive readjustment by flattening the cornea. There are different models of Intrastromal Corneal rings available: intrastromal corneal ring segments (ICRS) such as Keraring and intrastromal corneal continuous ring (ICCR) like Myoring.

Most studies of these two types of ring implantation outcomes are retrospective case series. Thus, this Randomized Clinical Trial study was designed with the aim of Comparing visual and refractive outcomes and complications of insertion Myoring versus Keraring using Femtosecond laser. Keratoconus patients with compound myopic astigmatism who meet the inclusion criteria will randomly allocated to the Keraring and Myoring groups. Subsequently, the clinical outcomes of two groups will be compared at one,3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* keratoconus patients and :
* age between 20 to 40
* corneal thickness> 380 microns
* mean keratometry between 44 to 60 D
* clear central cornea
* Patients should be discontinued their contact lenses for 3 weeks prior to the exams
* contact lenses in tolerance
* 20/200<visual acuity <20/30

Exclusion Criteria:

* Positive pregnancy test
* Breast-feeding
* History of glaucoma, cataract, vernal and atopic keratoconjunctivitis
* History of previous ophthalmologic surgery, keratorefractive surgery on the operative eye
* Dry eye
* Corneal stromal disorders
* History of herpetic keratitis
* Pellucid marginal degeneration
* Corneal grafts
* Retinal disorders
* Nystagmus and uncooperative disposition
* Neuro-ophthalmologic disorders
* Intraocular pressure <10 mmHg or >21 mmHg
* Patients with autoimmune, connective tissue disorders, diabetes and immunosuppressive drugs users
* Hyperopia

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Enrollment: 23
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
uncorrected visual acuity | 6 months
  Snellen E chart

SECONDARY OUTCOMES:
Corneal thickness | 6months
  Galilei Dual Scheimpflug Analyzer ( Ziemer, Switzerland)
Corneal irregularities (3, 5 and 7 mm of central cornea) | 6 months
  Galilei Dual Scheimpflug Analyzer ( Ziemer, Switzerland)
Front & back corneal elevation | 6 months
  Galilei Dual Scheimpflug Analyzer ( Ziemer, Switzerland)
Corneal aberrometry | 6 months
  Galilei Dual Scheimpflug Analyzer ( Ziemer, Switzerland)
Corneal eccentricity | 6 months
  Galilei Dual Scheimpflug Analyzer ( Ziemer, Switzerland)
Corneal hysteresis & corneal resistance factor | 6 months
  Ocular response Analyzer (reichert ophthalmic instruments, Buffalo,New York
  ,USA)
Intra and postoperative complications (glare, night vision problem, migration, extrusion, infection) | Intra and post operatien
  clinical examination, patients history

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Republic OF Iran, Tehran, Iran